CLINICAL TRIAL: NCT05109897
Title: Influencing Factors and Improving Strategy on Gait Variability in People With Parkinson's Disease
Brief Title: Influencing Factors on Gait Variability in PD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: 2021-08-014B
Record Dates: First submitted 2021-10-13; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease, Gait variability
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The principal motor features of Parkinson's disease (PD) include rigidity, tremor, bradykinesia, and postural instability. These motor deficits might cause gait dysfunction including reduced gait velocity, stride length, arm swing, and increased gait variability. Among these, increase in gait variability increased fall risk and served as a marker of disease progression. Previous studies reported that some factors might influence gait variability. However, which one contributes most has not yet been verified. Therefore, the purpose of the present study is to identify the more related influencing factors on gait variability in people with PD.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD
* Hoehn and Yahr stages I through III
* Ability to stand and walk 5 m independently with or without any walking aids
* Stable medication usage

Exclusion Criteria:

* Unstable medical conditions
* Any neurological, cardiopulmonary or orthopedic problem/diseases that may interfere with participating the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait variability | 10 minutes
  Using GAITRite system to measure coefficient of variation
Walking speed | 10 minutes
  Using GAITRite system to evaluate
Sensory organization test | 20 minutes
  Using NeuroCom Smart Balance Master to measure
Part III of the Unified Parkinson's Disease Rating Scale | 20 minutes
  The score ranged from 0 to 72. Higher scores show increased severity.
Tinetti Balance Scale | 10 minutes
  The score ranged from 0 to 28. Higher scores show better balance.
New freezing of gait questionnaire | 15 minutes
  The score ranged from 0 to 29. Higher scores show increased severity in freezing of gait.
Montreal Cognitive Assessment | 20 minutes
  The score ranged from 0 to 30. Higher scores show better cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided